CLINICAL TRIAL: NCT02820415
Title: Oocyte Accumulation by Vitrification is a Valid Strategy to Increase the Number of Euploid Available Embryos for Biopsy and Transfer After Preimplantation Genetic Testing
Brief Title: PGS on Blastocysts From Vitrified and Fresh Oocytes
Acronym: PGSvitfreov
Status: Completed | Type: Observational
Sponsor: Unità di Medicina della Riproduzione, Italy (Other)
Responsible Party: Principal Investigator, sandrine chamayou, Unità di Medicina della Riproduzione, Italy, Unità di Medicina della Riproduzione, Italy
Other Study IDs: Trial1
Record Dates: First submitted 2016-06-24; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Increase the Number of Blastocyst to Biopsy for Preimplantation Genetic Testing
Keywords: aneuploidy; next generation sequencing; oocyte vitrification; preimplantation genetic diagnosis; preimplantation genetic screening
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — DNA from trophectoderm cells

GROUPS / COHORTS (1):
- infertile couples undergoing ICSI for PGS/PGT: patients aged between 29.0 and 42.3 years, with basal FSH on day 3 between 2.9 and 12.0 IU/l. Undergoing 36 patients for RIF or RM. In each couple, the two partners had a normal karyotype. The patients underwent one to two cycles of ovarian stimulation to vitrify and accumulate oocytes and a last (second or third) cycle of ovarian stimulation. Ovarian stimulation was performed by the administration of recombinant FSH and LH (Gonal-F and Luveris: Merck-Serono, London, UK or Puregon, MSD, Franklin Lakes, USA) from cycle day 3 and luteal gonadotrophin-releasing hormone antagonist flexible schema (Cetrotide : Merck-Serono, London, UK).
  Interventions: Other: chromosomal status of blastocysts from fresh and vitrified/warmed oocytes

INTERVENTIONS:
Other: chromosomal status of blastocysts from fresh and vitrified/warmed oocytes

SUMMARY:
Oocyte accumulation by vitrification is a valid strategy to increase the number of available embryos for biopsy and the number of viable euploid embryos to transfer after preimplantation genetic testing.

DETAILED DESCRIPTION:
In the present study, the investigators considered the hypothesis to accumulate vitrified oocytes with a view to increasing the number of oocytes for micro-injection and consequently the number of blastocyst to diagnose for patients with normal ovarian reserve and candidate for PGT. The partecipants were proposed to undergo several cycles of ovarian stimulation. In the first cycles, mature (metaphase II) oocytes were vitrified and consequently accumulated. In the last cycle, the freshly produced mature oocytes and the previously accumulated ones were micro-injected together with the same partner's semen sample. PGT was performed on blastocysts produced from the two sources of oocytes. The comprehensive chromosomal analysis of biopsied trophectoderm cells was performed using NGS technology. The number of available euploid blastocyst and the proportion of euploid/aneuploidy embryos from fresh and vitrified/warmed oocytes were compared. In conclusion the investigators evaluated the efficacy of oocyte accumulation by vitrification in increasing the number of available embryos for biopsy and the number of viable euploid embryos to transfer after PGT.

ELIGIBILITY:
Inclusion Criteria:

* infertile women
* normal ovarian reserve
* with repeated implantation failure or reccurent miscarriage
* undergoing ICSI and asking to know the state of health of the embryos prior to embryo transfer

Ages: 28 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women, normal ovarian reserve, with repeated implantation failure or reccurent miscarriage
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
rate of euploidy in blastocyst from fresh and vitrified/warmed oocytes | 1 year
  from fresh and vitrified/warmed oocytes

CONTACTS AND LOCATIONS:
Locations (1):
- Sandrine Chamayou, Sant'Agata Li Battiati, Italy

REFERENCES:
- [Background] Chamayou S, Bonaventura G, Alecci C, Tibullo D, Di Raimondo F, Guglielmino A, Barcellona ML. Consequences of metaphase II oocyte cryopreservation on mRNA content. Cryobiology. 2011 Apr;62(2):130-4. doi: 10.1016/j.cryobiol.2011.01.014. Epub 2011 Jan 25. PMID 21272569
- [Background] Chamayou S, Alecci C, Ragolia C, Storaci G, Maglia E, Russo E, Guglielmino A. Comparison of in-vitro outcomes from cryopreserved oocytes and sibling fresh oocytes. Reprod Biomed Online. 2006 Jun;12(6):730-6. doi: 10.1016/s1472-6483(10)61085-1. PMID 16792849
- [Background] Chamayou S, Patrizio P, Storaci G, Tomaselli V, Alecci C, Ragolia C, Crescenzo C, Guglielmino A. The use of morphokinetic parameters to select all embryos with full capacity to implant. J Assist Reprod Genet. 2013 Jun;30(5):703-10. doi: 10.1007/s10815-013-9992-2. Epub 2013 Apr 13. PMID 23585186
- [Background] Chamayou S, Romano S, Alecci C, Storaci G, Ragolia C, Palagiano A, Guglielmino A. Oocyte vitrification modifies nucleolar remodeling and zygote kinetics-a sibling study. J Assist Reprod Genet. 2015 Apr;32(4):581-6. doi: 10.1007/s10815-015-0446-x. Epub 2015 Feb 21. PMID 25701142
- [Derived] Chamayou S, Sicali M, Alecci C, Ragolia C, Liprino A, Nibali D, Storaci G, Cardea A, Guglielmino A. The accumulation of vitrified oocytes is a strategy to increase the number of euploid available blastocysts for transfer after preimplantation genetic testing. J Assist Reprod Genet. 2017 Apr;34(4):479-486. doi: 10.1007/s10815-016-0868-0. Epub 2017 Jan 9. PMID 28070710